CLINICAL TRIAL: NCT05309174
Title: The Efficacy of Ultrasound Guided Superior Laryngeal Nerve Block as an Adjuvant to General Anesthesia During Vocal Cord Polypectomy by Laryngoscopy
Brief Title: The Study of Bilateral Upper Laryngeal Nerve Block for Supporting the Removal of Vocal Cord Polyps Under Laryngoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 789996
Record Dates: First submitted 2021-12-03; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Vocal Cord Polyp
Keywords: Ultrasound Guided Superior Laryngeal Nerve Block; Vocal Cord Polypectomy by Laryngoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia group (No Intervention): Patients received general anesthesia.
- General anesthesia combined laryngeal nerve block (Experimental): Group L received ultrasound-guided internal branch of the upper laryngeal nerve block (USG-guided iSLN block) bilaterally with 5 ml of 0.375% ropivacaine, along with general anesthesia.
  Interventions: Procedure: USG-guided iSLN block

INTERVENTIONS:
Procedure: USG-guided iSLN block — Ultrasound-guided internal branch of the upper laryngeal nerve block (USG-guided iSLN block) bilaterally with 5 ml of 0.375% ropivacaine , before general anesthesia.
  Arms: General anesthesia combined laryngeal nerve block

SUMMARY:
With the continuous development of microsurgery, supporting laryngoscopy acoustic polyp removal has become a very mature clinical operation. The operation has small trauma, short operation time, fast turnover and needing to wake up as soon as possible, but the supporting laryngoscopy has great stimulation to the throat and great hemodynamic fluctuations. This study aims to evaluate the efficacy of ultrasound guided superior laryngeal nerve block as an adjuvant to general anesthesia during vocal cord polypectomy by laryngoscopy.

DETAILED DESCRIPTION:
With the development of microsurgery, the vocal cord polypectomy by laryngoscopy has become a very mature surgery, under the laryngoscope. The surgery have some characteristics, that has a small trauma, shorter operative time, faster moving , but the strong stimulation of laryngeal surgery requires sufficient muscle relaxant condition, the greatest degree of reduce stress reaction, and waking up as soon as possible.

In the vocal cord polypectomy by laryngoscopy, the stimulation of throat often cause the nervous sympathetic excitement, including huge volatility in hemodynamics, fast heart rate, hypertension, cardiovascular serious adverse reactions such as ventricular arrhythmia, as placing the laryngoscope. Especially some patients are more obvious, who with a disease of hypertension, coronary atherosclerosis, tachycardia. It may cause myocardial ischemia and even other serious cardiovascular and cerebrovascular complications. In addition, it can also cause abnormal fluctuations in endocrine, immune and metabolism of the body, which has an important relationship with perioperative safety.

Superior laryngeal nerve block, blocking the laryngopharynx, epiglottis, tongue base, piriform recess and mucosa above the glottic fissure namely, can block the introduction of harmful stimuli and reduce pharyngeal stimulation during the perioperative period of endoscopic surgery. Bilateral superior laryngeal nerve block can reduce stress response effectively, maintaining hemodynamic stability, reducing perioperative adverse reactions and improving the safety of anesthesia. Furthermore, it can reduce the application of opioids and muscle relaxants during the operation, and shorten the time for patients to recover. Moreover, the vocal cords can be relaxed to provide good conditions for surgical operation. Accurate block of bilateral superior laryngeal nerve can also be used to provide good intraoperative and postoperative analgesia, under ultrasound guidance .

In this study, the anesthetic effect and patient status of general anesthesia and ultrasound guided superior laryngeal nerve block combined with general anesthesia were compared on the anesthesia of vocal cord polyp extraction under support laryngoscope.

The study method was to divide the subjects into experimental group and control group. The experimental group received ultrasound guided superior laryngeal nerve block combined with general anesthesia. However, the control group received all general anesthesia. The hemodynamic changes before endotracheal intubation (T1), during endotracheal intubation (T2), support laryngoscope placement (T3), immediately after extubation (T4), and 5minutes after extubation (T5) were recorded. The statistics of anesthetic dosage during operation were also recorded. Moreover, the investigators collect these results that the 9-item quality of recovery score (QOR-9) for 30 minutes and 60 minutes after extubation, the degree of cough immediately after extubation, 10 minutes, 1 hour and 4 hours after operation, and the degree of pharynx pain and hoarseness at 30 minutes, 2 hours, 4 hours and 24 hours after operation.

ELIGIBILITY:
Inclusion Criteria:

* To undergo direct rigid endoscopic laryngosurgery
* ASAⅠ～Ⅱ

Exclusion Criteria:

Coagulation disorders

* A history of neck surgery or an implant in the neck area
* Mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The degree of severity of sore-throat at just before extubation (bucking on the ETT) | At just before extubation (bucking on the ETT).
  Postoperative Sore-throat was assessed at just before extubation (bucking on the ETT) using a 4 grade scales. The degree of severity of sore throat is divided into four grades, grade 0: No sore throat, grade 1: Mild sore throat (complains of sore throat only upon inquiry) , grade 2: Moderate sore throat (complains of sore throat on his/her own), grade 3 :Severe sore throat (severe pain associated with marked change in voice).
The degree of severity of sore-throat at the time point of 10 minutes after extubation | At the time point of 10 minutes after extubation.
  Postoperative Sore-throat was assessed at 10 minutes after extubation using a 4 grade scales. The degree of severity of sore throat is divided into four grades, grade 0: No sore throat, grade 1: Mild sore throat (complains of sore throat only upon inquiry) , grade 2: Moderate sore throat (complains of sore throat on his/her own), grade 3 :Severe sore throat (severe pain associated with marked change in voice) .
The degree of severity of sore-throat at the time point of 1 hour after extubation | At the time point of 1 hour after extubation.
  Postoperative Sore-throat was assessed at 1 hour after extubation using a 4 grade scales. The degree of severity of sore throat is divided into four grades, grade 0: No sore throat, grade 1: Mild sore throat (complains of sore throat only upon inquiry) , grade 2: Moderate sore throat (complains of sore throat on his/her own), grade 3 :Severe sore throat (severe pain associated with marked change in voice) .
The degree of severity of sore-throat at the time point of 4 hour after extubation | At the time point of 4 hour after extubation.
  Postoperative Sore-throat was assessed at 1 hour after extubation using a 4 grade scales. The degree of severity of sore throat is divided into four grades, grade 0: No sore throat, grade 1: Mild sore throat (complains of sore throat only upon inquiry) , grade 2: Moderate sore throat (complains of sore throat on his/her own), grade 3 :Severe sore throat (severe pain associated with marked change in voice) .
The degree of severity of cough at the time point of 30 minutes following extubation | At the time point of 30 minutes following extubation.
  The degree of severity of cough is divided into four grades, grade 0: No cough, grade 1: Light or single cough, grade 2: Obvious to the observer, grade 3:Aphonia.
The degree of severity of cough at the time point of 2 hours following extubation | At the time point of 2 hours following extubation.
  The degree of severity of cough is divided into four grades, grade 0: No cough, grade 1: Light or single cough, grade 2: Obvious to the observer, grade 3:Aphonia.
The degree of severity of cough at the time point of 4 hours following extubation | At at the time point of 4 hours following extubation.
  The degree of severity of cough is divided into four grades, grade 0: No cough, grade 1: Light or single cough, grade 2: Obvious to the observer, grade 3:Aphonia.
The degree of severity of cough at the time point of 24 hours following extubation | At the time point of 24 hours following extubation.
  The degree of severity of cough is divided into four grades, grade 0: No cough, grade 1: Light or single cough, grade 2: Obvious to the observer, grade 3:Aphonia.
The degree of severity of hoarseness at the time point of 30 minutes following extubation. | At the time point of 30 minutes following extubation.
  The degree of hoarseness is divided into four grades, grade 0: None, grade 1:Noted by the patient, grade 2:More than one episode of unsustained (65 seconds) coughing, grade 3: Sustained (65 seconds) and Repetitive cough with head lift.
The degree of severity of hoarseness at the time point of 2 hours following extubation. | At the time point of 2 hours following extubation.
  The degree of hoarseness is divided into four grades, grade 0: None, grade 1:Noted by the patient, grade 2:More than one episode of unsustained (65 seconds) coughing, grade 3: Sustained (65 seconds) and Repetitive cough with head lift.
The degree of severity of hoarseness at the time point of 4 hours following extubation. | At the time points of 4 hours following extubation.
  The degree of hoarseness is divided into four grades, grade 0: None, grade 1:Noted by the patient, grade 2:More than one episode of unsustained (65 seconds) coughing, grade 3: Sustained (65 seconds) and Repetitive cough with head lift.
The degree of severity of hoarseness at the time point of 24 hours following extubation. | At the time point of 24 hours following extubation.
  The degree of hoarseness is divided into four grades, grade 0: None, grade 1:Noted by the patient, grade 2:More than one episode of unsustained (65 seconds) coughing, grade 3: Sustained (65 seconds) and Repetitive cough with head lift.

SECONDARY OUTCOMES:
Mean arterial pressure ( MAP) | Before endotracheal intubation (T1), during endotracheal intubation (T2), support laryngoscope placement (T3), immediately after extubation (T4), and 5 minutes after extubation (T5)
  Mean arterial pressure ( MAP) = Diastolic Pressure + 1 / 3 Pulse Pressure and normal value of 70~105 mmHg.
Heart rate (HR) | Before endotracheal intubation (T1), during endotracheal intubation (T2), support laryngoscope placement (T3), immediately after extubation (T4), and 5 minutes after extubation (T5)
  The heart rate range is 80-100 times / minutes, and the heart rate should be controlled in the normal range or ± 10%.
The 9-item quality of recovery score (QOR-9) | After extubation for 30 minutes and 60 minutes.
  The 9-item quality of recovery score is a validated scale with 5 domains. These measure physical comfort, emotional state, physical independence, psychological support, and pain. The minimum value is 0 and the maximum value is 18. Higher scores indicate better results
Anesthetic dosage | During operation
  The operative doses of remifentanil, and shufentanyl were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdi Yu, MD, Study Chair — Guizhou Provincial People's Hospital
Locations (1):
- Guizhou Provincial People's Hospital, Guiyang, Guizhou, China